CLINICAL TRIAL: NCT03125499
Title: A Prospective Observational Study to Evaluate Long-term Changes in Cartilage Morphology in Subjects Who Previously Received TPX-100 or Placebo in Study TPX-100-1 for Patellar Osteoarthritis Involving Both Knees
Status: Completed | Type: Observational
Sponsor: OrthoTrophix, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: TPX-100-4
Record Dates: First submitted 2017-04-11; First posted 2017-04-24 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Mild to Moderate Knee OA

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Previous treated with TPX-100 — No intervention, only observational
  Other Names: AC-100

SUMMARY:
To evaluate the long-term changes in patellar cartilage thickness in TPX-100 versus placebo-treated knees in subjects who participated in Study TPX-100-1 or TPX-100-2.

DETAILED DESCRIPTION:
No drug intervention. Study to collect 1 additional MRI of each knee treated in either TPX-100-1 or TPX-100-2.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who participated in TPX-100-1 and received 4 injections of 200 mg/injection TPX-100 in one knee, or subjects who participated in TPX-100
* Cruciate and collateral ligament stability as assessed by screening history and clinical examination
* Stable medial and lateral menisci as assessed by screening history and clinical examination
* Able to read, understand, sign and date the subject informed consent

Exclusion Criteria:

* Contraindication to MRI, including: metallic fragments, clips or devices in the brain, eye, or spinal canal; implanted devices that are magnetically programmed; weight > 300 lbs.; moderate or severe claustrophobia; previous intolerance of MRI procedure
* Prior surgery in the knees, excluding procedures for debridement only (no previous microfracture procedure)
* History of rheumatoid arthritis, psoriatic arthritis, or any other autoimmune or infectious cause for arthritis
* Last viscosupplementation (e.g. Synvisc® or similar hyaluronic acid product) injected into either knee < 3 months before enrollment
* Last intra-articular knee injection of corticosteroids < 3 months before enrollment
* Use of any steroids (except inhaled corticosteroids for allergy or respiratory problems) during the previous month before enrollment
* History of arthroscopy in either knee in the 3 months before enrollment
* History of septic arthritis, gout or pseudo-gout in either knee in the 12 months before enrollment
* Clinical signs of acute meniscal tear (locking, new acute mechanical symptoms consistent with meniscal tear)
* Active systemic infection
* Participation in other clinical osteoarthritis drug studies, except for studies TPX-100-1 and TPX-100-2, within two years prior to enrollment in TPX-100-4.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with bi-lateral knee OA that have previous been treated in TPX-100-1 or TPX-100-2
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the long-term changes in patellar cartilage thickness | Between 24 and 34 months from initial drug treatment
  Quantitative analysis of long-term changes in patellar cartilage thickness by MRI

SECONDARY OUTCOMES:
Examine intra-subject longitudinal changes in patellar cartilage volume between TPX-100 versus placebo-treated knees by MRI | Between 24 and 34 months from initial drug treatment
  Examine intra-subject longitudinal changes in patellar cartilage volume between TPX-100 versus placebo-treated knees by MRI
Examine intra-subject longitudinal changes in thickness and thinness scores of cartilage in the central (non-patellar) compartment of knees | Between 24 and 34 months from initial drug treatment
  Examine intra-subject longitudinal changes in thickness and thinness scores of cartilage in the central (non-patellar) compartment of knees
Examine intra-subject longitudinal changes in Patient reported outcome measures | Between 24 and 34 months from initial drug treatment
  Examine intra-subject longitudinal changes in Patient Reported Outcome Measures

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Samy Metyas, Covina, California, United States

IPD SHARING:
Plan to Share IPD: No